CLINICAL TRIAL: NCT02375022
Title: A Study to Evaluate the Efficacy of Rh-Endostatin (Endostar®) in Combination With Icotinib for Advanced Non-Small Cell Lung Cancer With EGFR Mutations
Brief Title: Rh-Endostatin in Combination With Icotinib for Advanced NSCLC With EGFR Mutations
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Zhejiang University (Other)
Collaborators: Jiangsu Simcere Pharmaceutical Co., Ltd. (Industry); Beta Pharma, Inc. (Industry)
Responsible Party: Principal Investigator, Qiong Zhao, Chief, Department of Thoracic Oncology, Zhejiang University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ZYTOP1501
Record Dates: First submitted 2015-02-10; First posted 2015-03-02 (Estimated); Last update posted 2015-03-24 (Estimated); Status verified 2015-03

CONDITIONS: Lung Cancer
MeSH Terms: conditions — Lung Neoplasms | interventions — endostar protein; icotinib; Endostatins

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Endostar and icotinib (Experimental): Combination of drug: Endostar: 15mg CIV d1-9, Q3w and icotinib: 125mg TID po. If no progressive disease observed, combination treatment will continue until unacceptable toxicity or progressive disease.
  Interventions: Drug: Endostar and icotinib

INTERVENTIONS:
Drug: Endostar and icotinib — Endostar and icotinib are used as combination therapy.
  Other Names: Recombinant Human Endostatin Injection; Icotinib Hydrochloride Tablets

SUMMARY:
This single-arm pilot study tries to invesitgate how well giving icotinib with rh-endostatin (Endostar®) works in treating patients with advanced stage non-small cell lung cancer (NSCLC) with epidermal growth factor receptor (EGFR) activating mutations. Icotinib may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth. Anti-angiogeneiss drug, such as rh-endostatin, can block tumor growth by inhibiting the ability of tumors to grow new blood vessels and spread. It is not yet known whether icotinib is more effective when given with rh-endostatin in NSCLC patients with EGFR activating mutations.

DETAILED DESCRIPTION:
1. Open-label, single-arm, prospective pilot study.
2. Definition of advanced non small cell lung cancer: stage IIIb or IV. EGFR mutation status: activating mutation (defined as deletion 19 or exon 21 L858R mutation).
3. Before starting study treatment, computed tomography scans of the chest, B ultrasound of abdomen, 12-lead electrocardiogram, MRI scan of brain, and a bone scan are required.
4. Tumor response, based on investigator-assessed Response Evaluation Criteria in Solid Tumors (RECIST v.1.1), will be evaluated every 6 weeks during treatment.
5. Exploratory evaluation will be performed using dynamic contrast enhanced MRI (DCE-MRI).
6. QoL will be assessed using the core module, which will be completed by patients at baseline and before each cycle during treatment.
7. All patients who prematurely discontinue treatment for any reason will be followed for survival.

ELIGIBILITY:
Inclusion Criteria:

* Histologic documentation of non small cell lung cancer, with activating epidermal growth factor receptor (defined as deletion 19 or exon 21 L858R mutation).
* Stage IV disease according to the 7th Edition of the American Joint Committee on Cancer staging system -Measureable disease
* Life expectancy of >= 12 months
* Eastern Cooperative Oncology Group (ECOG) Performance Status (PS) 0 or 1
* Absolute neutrophil count (ANC) >= 1, 500/mm^3, platelet count >= 100,000/mm^3, hemoglobin >= 9.0 g/dL.
* Total bilirubin =< 1.5 x upper limit of normal (ULN), serum glutamic oxaloacetic transaminase (SGOT) (aspartate aminotransferase [AST]) and serum glutamic pyruvic transaminase (SGPT) (alanine aminotransferase [ALT]) =< 2.5 x ULN in patients without liver or bone metastases; < 5 x ULN in patients with liver or bone metastases, cockcroft-Gault calculated creatinine clearance of >= 45 ml/min or creatinine =< 1.5 x ULN.
* Prothrombin time (PT) =< 1.5 x ULN, partial thromboplastin time (PTT) =< ULN
* Urine dipstick proteinuria < 2+. Patients discovered to have >= 2 + proteinuria on dipstick urinalysis at baseline should undergo a 24-hour urine collection and must demonstrate < 1 g of protein in 24 hours.
* Negative pregnancy test done =< 7 days prior to randomization, for women of childbearing potential only.
* Provide informed written consent.
* Willing to return to enrolling institution for follow-up.
* Willing to provide tissue and blood samples for correlative research purposes.

Exclusion Criteria:

* Evidence of bleeding diathesis or coagulopathy.
* Evidence of central nervous system involvement or brain metastases confirmed by head CT or brain MRI within 28 days prior to being registered for protocol therapy.
* Major surgical procedure, open biopsy, or significant traumatic injury within 28 days prior to registration for protocol therapy.
* Anticipation of need for major surgical procedure during the course of the study.
* Minor surgical procedures such as fine needle aspirations or core biopsies within 7 days prior to registration for protocol therapy.
* History of abdominal fistula, gastrointestinal perforation, or intra-abdominal abscess within 6 months prior to registration for protocol therapy.
* Serious, non-healing wound, ulcer, or bone fracture.
* History of hemoptysis.
* Clinically significant infections as judged by the treating investigator.
* Other active malignancy

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2015-03; Primary Completion 2016-03 (Estimated); Study Completion 2016-03 (Estimated)

PRIMARY OUTCOMES:
Objective response rate | 6 months

SECONDARY OUTCOMES:
Progression free survival | 12 months
Safety: Number of Participants with Adverse Events | 12 months
  Number of Participants with Adverse Events as a Measure of Safety and Tolerability

CONTACTS AND LOCATIONS:
Locations (1):
- Zhejiang University, Hangzhou, Zhejiang, China